CLINICAL TRIAL: NCT05214391
Title: Safety and Efficacy of Zanubrutinib in the Treatment of Immune Thrombocytopenia
Brief Title: A Prospective, One-arm and Open Clinical Study of Zanubrutinib in the Treatment of Immune Thrombocytopenia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2021047
Record Dates: First submitted 2022-01-19; First posted 2022-01-28 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-01

CONDITIONS: Immune Thrombocytopenia; Treatment
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — zanubrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Intervention ( zanubrutinib) (Experimental): 30 enrolled patients are picked up to take zanubrutinib at the indicated dose.
  Interventions: Drug: Zanubrutinib

INTERVENTIONS:
Drug: Zanubrutinib — The initial dose is 80mg/day. If the treatment is ineffective after 4 weeks, and under the condition of good safety, the investigator will judge that the dosage should be added to 80mg twice/day，or a higher dose for oral maintenance. The maximum dose is 160mg twice a day. The duration of zanubrutinib is 24 weeks.
  In case of intolerable adverse reactions, such as severe infection, severe bleeding, hematopenia, arrhythmia, etc., investigator can reduce the dose of zanubrutinib, or withdraw from clinical trials as appropriate.
  Other Names: The treatment of zanubrutinib

SUMMARY:
To evaluate the safety and efficacy of zanubrutinib in the treatment of immune thrombocytopenia in 30 patients.

DETAILED DESCRIPTION:
Immune thrombocytopenia (ITP) is an organ-specific autoimmune disease, which is characterized by decreased platelet count and skin and mucosal bleeding. ITP is a kind of disease with increased platelet destruction and impaired platelet production caused by autoimmunity. Conventional treatment of adult ITP includes first-line glucocorticoid and immunoglobulin therapy, second-line TPO and TPO receptor agonist, splenectomy and other immunosuppressive treatments (such as rituximab, vincristine, azathioprine, etc.). ITP is one of the most common hemorrhagic diseases. At present, the treatment response of ITP is not good, and a considerable number of patients need drug maintenance treatment, which seriously affects the quality of life of patients and increases the economic burden of patients. Therefore, there is still a lack of effective treatment for adult ITP, especially for refractory ITP patients, which is one of the problems that have attracted more attention and need to be solved urgently.

BTK inhibitors can affect autoimmune diseases (AID) involving B cells and non-B cells through B cell receptor, Fc receptor and RANK receptor signals, such as systemic lupus erythematosus (SLE), multiple sclerosis (MS) and rheumatoid arthritis (RA) .Therefore, small molecule BTK inhibitors can treat autoimmune diseases by targeting B cells. At present, clinical studies on the treatment of immune thrombocytopenia with BTK inhibitor (BRN1008) have been carried out abroad. The preliminary results show that 50% of patients in the treatment ≥ 12 weeks and the initial dose is 400 mg BID group have reached the primary endpoint and maintained platelet response.

Zebutinib is a new selective Bruton tyrosine kinase (BTK) inhibitor developed by Baekje Shenzhou Company of China. In November 2019, it was approved by the US Food and Drug Administration to treat adult mantle cell lymphoma (MCL) patients who had received at least one treatment before. Compared with the first generation BTK inhibitors (ibutinib and acalabrutinib), zebutinib has stronger targeting and fewer adverse reactions.

Therefore, the investigators designed this clinical trial to provide new treatment options for clinical treatment of ITP.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and above, male or female；
* Conform to the diagnostic criteria of immune Thrombocytopenia (ITP)；
* Diagnosis of ITP>3 months；
* Primary ITP with a platelet count of <30 X 109/L prior to inclusion with failure to achieve response or relapse after corticosteroid therapy, and at least one second-line therapy including rituximab >12 weeks ago and/or TPO-RAs.
* Liver and kidney function, such as ALT, AST, BUN, SCR < 1.5 × upper limit of normal value, passing physical examination;
* ECOG physical state score ≤ 2 points；
* Cardiac function of the New York Society of Cardiac Function ≤ 2；
* Signed and dated written informed consent.

Exclusion Criteria:

* Uncontrollable primary diseases of important organs, such as malignant tumors, liver failure, heart failure, renal failure and other diseases;
* HIV positive;
* Accompanied by uncontrollable active infection, including hepatitis B, hepatitis C, cytomegalovirus, EB virus and syphilis positive;
* Accompanied by extensive and severe bleeding, such as hemoptysis, upper gastrointestinal hemorrhage, intracranial hemorrhage, etc.;
* At present, there are heart diseases, arrhythmias that need treatment or hypertension that researchers judge is poorly controlled;
* Patients with thrombotic diseases such as pulmonary embolism, thrombosis and atherosclerosis;
* Those who have received allogeneic stem cell transplantation or organ transplantation in the past;
* Patients with mental disorders who cannot normally obtain informed consent and conduct trials and follow-up;
* Patients whose toxic symptoms caused by pre-trial treatment have not disappeared;
* Other serious diseases that may limit the subject's participation in this test (such as diabetes; Severe cardiac insufficiency; Myocardial obstruction or unstable arrhythmia or unstable angina pectoris in recent 6 months; Gastric ulcer, etc.);
* Patients with septicemia or other irregular severe bleeding;
* Patients taking antiplatelet drugs at the same time;
* Pregnant women, suspected pregnancies (positive pregnancy test for human chorionic gonadotropin in urine at screening) and lactating patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-02-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with a platelet count ≥ 30 × 10^9/L and 50×10^9/L at week 12(Day 85) | 12 weeks
  Observe the changes of blood routine platelet count after 12 weeks of treatment, and calculate the proportion and times of subjects ≥ 30 × 10^9/L and 50 × 10^9/L.

SECONDARY OUTCOMES:
Persistent platelet response with clinical significance at 24 weeks | 24 weeks
  Response defined as as the proportion of subjects with platelet count ≥ 50 × 109/L in at least 4 of the last 6 visits within 24 weeks without rescue treatment.
Number of participants with clinically significant bleeding as assessed using the world health organization (WHO) bleeding scale. | 24 weeks
  The WHO Bleeding Scale is a measure of bleeding severity with the following grades: grade 0 = no bleeding, grade 1= petechiae, grade 2= mild blood loss, grade 3 = gross blood loss, and grade 4 = debilitating blood loss.
The occurrence of adverse events during treatment (AE/SAE), treatment-related adverse events (TRAE) and serious adverse events (TRSAE) | 24 weeks
  The occurrence of adverse events during treatment (AE/SAE), treatment-related adverse events (TRAE) and serious adverse events (TRSAE)
Measurements of antibodies and various subsets of immunocompetent cells | 24 weeks
  Changes of anti-GPIIb/IIIa and Ib antibody and and various subsets of immunocompetent cells during study

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zhang, MD, Principal Investigator — Chinese Academy of Medical Science and Blood Disease Hospital
Locations (1):
- Chinese Academy of Medical Science and Blood Disease Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Researchers qualified can request the dataset, including de-identified individual subject data. Data may be requested from PI from 12 months 36 months after study completion.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 12 months to 36 months after study completion
Access Criteria: Upon request to PI.